CLINICAL TRIAL: NCT01899313
Title: A Cognitive Behavioral Therapy-Based Text Message Intervention for Methamphetamine Dependence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: California Pacific Medical Center Research Institute (Other)
Responsible Party: Principal Investigator, Gantt Galloway, PharmD, Senior Scientist, California Pacific Medical Center Research Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2012.119-2
Record Dates: First submitted 2013-05-30; First posted 2013-07-15 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Amphetamine-Related Disorders
Keywords: methamphetamine dependence; texting; short message service; addiction; amphetamine; outpatient
MeSH Terms: conditions — Amphetamine-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT- based SMS text messaging intervention (Experimental): cognitive behavioral therapy- (CBT-) based short message service (SMS) text messaging intervention
  Interventions: Behavioral: CBT- based SMS text messaging intervention; Behavioral: CBT group therapy
- Placebo Texts (Placebo Comparator): Placebo texts will be given instead of interventional texts
  Interventions: Behavioral: CBT group therapy

INTERVENTIONS:
Behavioral: CBT- based SMS text messaging intervention
  Arms: CBT- based SMS text messaging intervention
Behavioral: CBT group therapy
  Other Names: Cognitive Behavioral Group Therapy

SUMMARY:
This Phase I behavior therapy development study seeks to improve treatment outcomes for methamphetamine (MA)-dependent subjects by developing a novel cognitive behavioral therapy- (CBT-) based short message service (SMS) text messaging intervention.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults ≥ 18 years who are seeking treatment for MA addiction.
* Own a cellular phone with SMS text messaging capability and have an unlimited text messaging plan.
* Available to attend CBT therapy groups.
* Agreeable to conditions of the study and signed an informed consent form.

Exclusion Criteria:

* Projected to be unavailable > 12 hours/day to read and send text messages.
* Any medical or psychosocial condition that would preclude safe, useful, or consistent participation,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of MA-negative urine samples between the 2-week CBT text period and the 2-week control period | 5 weeks
  The primary efficacy measure for this study is the difference in proportion of MA-negative urine samples between the 2-week CBT text period and the 2-week control period. Urine samples will be analyzed for MA by immunoassay with a cutoff of 1,000 ng/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Gantt Galloway, PharmD, Principal Investigator — California Pacific Medical Center
Locations (2):
- United States (2):
  - New Leaf Treatment Center, Lafayette, California
  - Addiction & Pharmacology Research Laboratory, San Francisco, California

REFERENCES:
- See also: clinical site at which patients are seen — http://nltc.com/